CLINICAL TRIAL: NCT06321978
Title: Observational Study to Describe the Utilization of Foam Dressings in Routine Clinical Practice, for the Treatment of Patients With Chronic Wounds in Primary Healthcare Centers in Spain.
Brief Title: Mepilex Border Flex Utilization Pilot Spain
Acronym: MxBFlexUPESP
Status: Recruiting | Type: Observational
Sponsor: Molnlycke Health Care AB (Industry)
Responsible Party: Sponsor
Other Study IDs: MxBFlexUP ESP
Record Dates: First submitted 2024-02-29; First posted 2024-03-20 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Wound
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other

GROUPS / COHORTS (1):
- Study Group: Mepilex Border Flex dressing changes
  Interventions: Device: Mepilex Border Flex

INTERVENTIONS:
Device: Mepilex Border Flex — Usage of Mepilex Border Flex according to intended use and standard of care.

SUMMARY:
The aim of this study is to assess and describe the utilization of Mepilex® Border Flex and other foam dressings available in routine clinical practice in the management of patients with chronic wounds, in order to understand the pattern of use and the frequency of dressing changes in wound management. The study will also allow to gain information about the opinion of the HCPs and the patient's experience concerning wound management with foam dressings. This information may help to understand patient's health care optimization in terms of quality and efficiency.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older.
* The patient has been deemed by the HCP to change dressing to Mepilex® Border Flex.
* Patients with chronic wounds (wounds that have not reduced in size by more than 40% to 50% or healed within a month) treated with foam dressings, other that Mepilex® Border Flex, according to its intended use at baseline visit for minimum 4 weeks.
* Patients with an expectation of wound follow-up of at least 4 weeks.
* Patients agree only to have the dressing changed by the HCP.
* Patients capable of signing the Informed Consent Form and answer the questions being asked.

Exclusion Criteria:

* Patients with any applicable contraindication or sensibilization to any of the dressing compounds
* Patients with pressure ulcers (PU) stage I, deep tissue injuries or terminal wounds (e.g., fungating wounds)
* Patients with wounds whose location and/or aetiology requires a dressing change for reasons that are unrelated to the dressing characteristics such as wounds in the sacral area.
* Hospice patients
* Patients participating in other studies interfering with this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is addressed to adult patients with chronic wounds- wounds that have not reduced in size by more than 40% to 50% or healed within a month, and who are already being treated with a foam dressing. The patient must be deemed by HPC to be treated with Mepilex® Border Flex according to the indications of the dressing.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-02-16 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Dressing use | 4 weeks
  Number of dressings used the week before baseline visit compared to the number of dressings used the week before follow-up visit.

SECONDARY OUTCOMES:
Wound characteristics | 4 weeks
  Describe clinical characteristics of chronic wounds that are treated with foam dressings in routine clinical practice by HCP assessment
Wound management | 4 weeks
  Describe the management of chronic wounds in terms of frequency of dressing change, type of dressings used and reason for dressing change
Technical Performance (HCP evaluation) | 4 weeks
  Several questions will be asked to evaluate the technical performance properties of the primary dressing. The following will be assessed by the investigator/designee using no/yes values:
  1) Based on this patient, would you recommend Mepilex Border Flex for use in your organisation?
  All other properties will be assessed by the investigator/designee using a 3-item scale of worse, same, better. These include:
  * Ease of application
  * Ease of removal
  * Ability to conform to wound site
  * Ability to indicate the need for dressing change
  * Ability to stay in place
  * Trauma to the wound bed
  * Ability to indicate the need for dressing change
  * Trauma to the wound bed
  * Trauma to the peri-wound skin
  * Patient concordance
  * Overall dressing performance
Patient Experience (PRO) | 4 weeks
  Patients are asked to rate the dressings in regards their experience
  The following questions will be assessed by the investigator/designee using a 1-10 level visual analogue scale for pain:
  * How wound you rate the pain in your wound today?
  * How would you rate the pain when Mepilex Border Flex was removed from your wound today?
  The following will be assessed by the investigator/designee using no/yes values:
  *Would you recommend this treatment to a relative or friend?
  All other properties will be assessed by the investigator/designee using a 4-item scale of very poor, poor, good, very good. These include:
  * How would you rate the comfort of Mepilex Border Flex applied to your wound?
  * How would you rate Mepilex Border Flex used in regards to the ability to stay in place?
  * How would you rate your overall satisfaction regarding wound management (including the properties of Mepilex Border Flex and treatment of your wound)
Costs | 4 weeks
  Estimate the weekly cost per patient associated with the dressings used in wound care episodes and the characteristics of use by evaluating type and size of wound and frequency of dressing change

CONTACTS AND LOCATIONS:
Locations (1):
- CS Ciudad Expo - Mairena de Aljarafe, Seville, Andalusia, Spain